CLINICAL TRIAL: NCT05501132
Title: Efficacy of Transcranial Direct Current Stimulation (tDCS) in Symptoms, Quality of Life, Cognitive Deficits and Brain Physiology of Patients with Obsessive-compulsive Disorder
Brief Title: Efficacy of Intensified Transcranial Direct Current Stimulation in Obsessive-compulsive Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The National Brain Mapping Laboratory (NBML) (Other)
Collaborators: Ardabil University of Medical Sciences (Other); Leibniz Research Centre for Working Environment and Human Factors (Other)
Responsible Party: Principal Investigator, Mohammad Ali Salehinejad, Principal Investigator, Technical University of Dortmund
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IR.ARUMS.REC.1399.102
Record Dates: First submitted 2022-08-12; First posted 2022-08-15 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2023-11

CONDITIONS: Obsessive-Compulsive Symptom
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- tDCS group 1 (Experimental): In the first experimental group, the TDCS intervention protocol consists of 10 sessions of 20 minutes of 1 mA electrical stimulation on 5 consecutive days with two sessions per day.
  Interventions: Device: transcranial direct current stimulation
- tDCS group 2 (Experimental): In the second experimental group, the TDCS intervention protocol consists of 10 sessions of 20 minutes of 2 mA electrical stimulation on 5 consecutive days with two sessions per day.
  Interventions: Device: transcranial direct current stimulation
- Control group (Placebo Comparator): In the placebo group, the TDCS intervention protocol consists of 10 sessions of 20 minutes of sham electrical stimulation on 5 consecutive days with two sessions per day.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — Patients will receive 10 sessions of 20 minutes of either 1 mA, 2 mA or sham electrical stimulation on 5 consecutive days
  Other Names: tDCS

SUMMARY:
This is a randomized, double-blind, parallel-group, sham-controlled trial that aims to investigate the effectiveness of transcranial direct current stimulation (TDCS) on improving symptoms, quality of life, depression, and cognitive functions in 39 patients with obsessive-compulsive disorder (OCD) that are randomized in 3 experimental groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Obsessive-compulsive Disorder by a psychiatrist and DSM-5-based behavioral checklist
* being 18-50 years old
* providing written informed consent
* If female, negative urine pregnancy test
* stable medication regime especially the classical neuroleptics and all CNS-activating medications, if taken, 4-6 weeks before the experiment and during the experiment

Exclusion Criteria:

* smoker
* pregnancy
* alcohol or substance dependence
* history of seizure
* history of neurological disorder
* history of head injury
* presence of ferromagnetic objects in the body that are contraindicated for brain stimulation of the head (pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips, metallic prostheses, permanent eyeliner, implanted delivery pump, or shrapnel fragments) or fear of enclosed spaces.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Yale-Brown Obsessive-Compulsive (Y-BOCS) rating scale | up to 1 month after the intervention
  Score in the Yale-Brown Obsessive-Compulsive (Y-BOCS). Total scores on the measure range from 0 to 40, with a score of 0-7 indicating subclinical symptoms, 8-15 mild symptoms, 16-23 moderate symptoms, 24-31 severe symptoms and 32-40 extreme symptoms.
Beck Anxiety Questionnaire (BAI) | up to 1 month after the intervention
  Score in the Beck Anxiety Questionnaire (BAI). The BAI scores are classified as minimal anxiety (0 to 7), mild anxiety (8 to 15), moderate anxiety (16 to 25), and severe anxiety (30 to 63).
Response inhibition task 1 | up to 1 month after the intervention
  Performance in the response inhibition tasks (Flanker test)
Working memory task | up to 1 month after the intervention
  Performance in the working memory task as an executive function task
Response inhibition task 2 | up to 1 month after the intervention
  Performance in the response inhibition tasks (Go/No-Go task)

SECONDARY OUTCOMES:
Beck Depression Questionnaire (BDI-II) | up to 1 month after the intervention
  Score in the Beck Depression Questionnaire (BDI-II). The BDI-II scores are classified as below:
  Score of 1-10: These ups and downs are considered normal. Score of 11-16: Mild mood disturbance. Score of 17-20: Borderline clinical depression. Score of 21-30: Moderate depression. Score of 31-40: Severe depression. Score of 40+ Extreme depression.
Quality of Life Questionnaire (WHOQUL) | up to 1 month after the intervention
  Score in the Quality of Life Questionnaire. It has 26 items and each item is rated on a 5-point scale with a higher score indicative of higher quality of life.
electroencephalogram (EEG) oscillatory power | up to 1 month after the intervention
  Change in the EEG power in alpha, delta, theta and beta bands
electroencephalogram (EEG) functional connectivity | up to 1 month after the intervention
  Change in the EEG functional connectivity

CONTACTS AND LOCATIONS:
Locations (1):
- Ardabil University of Medical Sciences, Ardabil, Iran

IPD SHARING:
Plan to Share IPD: No